CLINICAL TRIAL: NCT02970929
Title: A 26-Week Open-label Safety and Tolerability Extension Study of SEP-363856 in Adult Subjects With Schizophrenia
Brief Title: An Extension Study of Safety and Tolerability of SEP-363856 in Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-202; 2016-001556-21 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental): SEP-363856 capsule (25 mg, 50 mg, or 75 mg) once daily
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — One SEP-363856 capsule (25 mg, 50 mg or 75 mg (flex)) daily for 26 weeks

SUMMARY:
An extension study of safety and tolerability of SEP-363856 in adult subjects with schizophrenia

DETAILED DESCRIPTION:
This is a 26 week, multiregional, open-label extension study designed to evaluate the long-term safety and tolerability of SEP-363856 for the treatment of subjects with schizophrenia who have completed the 4 week double-blind treatment phase of Study SEP361-201 (NCT02969382) Subjects received open-label SEP-363856 50 mg/day from Day 1 through Day 3, and then received flexible dosing of SEP-363856 (25, 50, or 75 mg/day) for the rest of the trial.

No statistical hypothesis tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

Subject must give written informed consent and privacy authorization prior to participation in the study and able to comply with the protocol, in the opinion of the investigator.

* Subject has completed Study SEP361 201 through Week 4
* Subject has not taken any medication other than the study drug for the purpose of controlling schizophrenia symptoms during Study SEP361 201.
* Female subject must have a negative urine pregnancy test at Visit 7 of Study SEP361 201; females who are post-menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Male subjects with female partner(s) of childbearing potential must agree to avoid fathering a child and use acceptable methods of birth control from screening until at least 30 days after the last study drug administration

Exclusion Criteria:

* Subject answers "yes" to "suicidal ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at Visit 7 of Study SEP361 201. Subjects who answer "yes" to this question must be referred to the Investigator for follow up evaluation.
* Subject has a clinically significant abnormality including physical examination, vital signs, ECG, or laboratory test at Visit 7 of Study SEP361 201 that the investigator in consultation with the medical monitor considers to be inappropriate to allow participation in the study.
* Subject has a positive urine drug screen (UDS) or breath alcohol test at Visit 7 of Study SEP361 201.
* Subject is pregnant or lactating.
* Subject is at high risk of non-compliance in the Investigator's opinion.
* Subject is in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (6):
  - Woodland International research Group, Little Rock, Arkansas
  - CNRI-Los Angeles, LLC, Pico Rivera, California
  - UCSD Medical Center UCSD Department of Psychiatry, San Diego, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Kashinath Yadalam, Lake Charles, Louisiana
  - Pillar Clinical Research, LLC, Dallas, Texas
- Hungary (2):
  - Bugát Pál Kórház-Rendelőintézet, Rehabilitációs Elmegyógyászati Osztály, Gyöngyös, Dózsa György
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Pszichiatriai Osztaly, Gyula
- Romania (4):
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Centrul de Evaluarea si Tratament al Toxicodependentelor pentru Tineri "Sf. Stelian", Sectia Psihiatrie, Bucharest
  - spitalul Clinic de Neuropsihiatrie Craiova ,Clinica II Psihiatrie, Craiova
  - Institutul de Psihiatrie Socola Iasi, Sectia Psihiatrie III Acuti, Iași
- Russia (8):
  - St-Petersburg SHI Psychiatrical hospital #1 n.a. Kaschenko, Gatchina
  - City Psychiatric Hospital of St. Nikolay Chudotvorets, Saint Petersburg
  - FB=SBI"Saint Petersburg Scientific and Research Psychoneurological Institute n.a. V.M. Bekhterev", Saint Petersburg
  - SPHI "City Mental Hospital #3 n.a. I.I.Skvortsov-Stepanov", Saint Petersburg
  - SPb SBIH "City Psychoneurological Dispensary #7 (with inpatient facilities)", Saint Petersburg
  - SHI Regional Clinical Psychiatry Hospital of St. Sofia, Saratov
  - FSBEI HE "Smolensk State Medical University" of the MoH of the RF, Smolensk
  - Sverdlov Regional Psychiatric Clinical Hospital, Yekaterinburg
- Ukraine (10):
  - Regional Psychoneurological Hospital #3, Dept of Crisis Cond & Primary Psych Episode #1, Ivano-Frankivsk
  - CHI Kharkiv RCPH#3 Center of Emerg PsychSI Inst of Neur, Psych & Narc of NAMSU, Unit of Emergency Psychiatry and Narcology, Kharkiv
  - CHI Kharkiv Regional Clinical Psychiatric Hospital #3, Psychiatric Department of Primary Psychotic Episod, Kharkiv
  - CI Kherson Regional Psychiatric Hospital of Kherson RC, Kherson
  - TMA Psychiatry in Kyiv Center of NT & Rehabilitation of Psychotic Conditions, Kyiv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - CI Cherkasy Regional Psychiatric Hospital of ChRC, Femail Dept #11, Male Dept #12, Smila
  - Ternopil RCCPH Depts of Psychiatry #2 (m) & Psychiatry #6 Ternopil I.ya. Gorbachevskyi SMU, Ternopil
  - Transcarpathian Regional Narcological Dispensary, Uzhhorod
  - CI O.I. Yuschenko VRPsH Depts #7 & #10 M.I. Pyrogov VNMU, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received open-label SEP-363856 50 mg/day from Day 1 through Day 3, and then received flexible dosing of SEP-363856 (25, 50, or 75 mg/day) for the rest of the trial.
Period: Overall Study
Arm/Group | SEP-363856
Started | 157
Subjects Who Received Study Medication | 156
Completed | 105
Not Completed | 52
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 8
Not completed — NON-COMPLIANCE WITH STUDY DRUG | 1
Not completed — INVESTIGATOR CONSIDERS SUBJECT CLINICALLY UNSTABLE, NOT APPROPRIATE FOR DISCHARGE TO AN OUTPATIENT | 1
Not completed — SPONSOR REQUEST THAT SUBJECT BE WITHDRAWN DUE TO POSITIVE DRUG RESULTS AND FOR THE SUBJECT'S SAFETY | 1
Not completed — LOST TO FOLLOWUP | 6
Not completed — MOVED OUT OF STATE | 1
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 154
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 151
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 136
  More than one race | 1
  Unknown or Not Reported | 0
Age, Customized [Count of Participants; unit: Participants]
  >=18 - <25 years | 38
  >=25 - <=40 years | 118
Country [Count of Participants; unit: Participants]
  Hungary | 8
  Romania | 6
  Russia | 68
  Ukraine | 54
  United States | 20
Double-blind Baseline BMI (Body Mass Index) Group [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 2
  >=18.5 - <25.0 kg/m^2 | 80
  >=25.0 - <30.0 kg/m^2 | 55
  >=30.0 kg/m^2 | 19
Open-label Baseline BMI (Body Mass Index) Group [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 3
  >=18.5 - <25.0 kg/m^2 | 82
  >=25.0 - <30.0 kg/m^2 | 53
  >=30.0 kg/m^2 | 18
Open-label Baseline Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 85.20 (13.467)
Open-label Baseline BMI (Body Mass Index) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.05 (3.890)
Open-label Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 75.32 (13.987)
Open-label Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 173.1 (7.73)
Double-blind Baseline Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 85.36 (13.508)
Double-blind Baseline BMI (Body Mass Index) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.07 (3.863)
Double-blind Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 75.38 (13.873)
Double-blind Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 173.1 (7.73)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Overall Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events (AEs) Leading to Discontinuation
Description: Number of Participants with overall Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events (AEs) leading to discontinuation
Time Frame: From first dose of study drug to last study visit (27 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Participants
  Overall Adverse Events (AEs) | 88
  Serious Adverse Events (SAEs) | 15
  Adverse Events leading to discontinuation from study | 18
  Adverse Events leading to discontinuation of study drug | 18

2. Secondary Outcome: Frequency of Suicidal Ideation (SI) and Suicidal Behavior (SB) Using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: Number of participants with suicidal ideation (SI) and suicidal behavior (SB) using the Columbia - Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a tool designed to systematically assess and track suicidal behavior and suicidal ideation for life time, one month prior to the screening visit for suicidal ideation and 6 months prior to the screening visit for suicidal behavior, and throughout the study. The strength of this suicide classification system is in its ability to comprehensively identify suicidal events while limiting the over-identification of suicidal behavior.
Time Frame: Overall post Open-label Baseline treatment period (26 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Participants
  Any suicidal ideation | 3
  Any suicidal behavior | 1
  Any suicidality | 3

3. Secondary Outcome: Severity of Suicidal Ideation (SI) and Suicidal Behavior (SB) Using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a tool designed to systematically assess and track suicidal behavior and suicidal ideation for life time, one month prior to the screening visit for suicidal ideation and 6 months prior to the screening visit for suicidal behavior, and throughout the study. The strength of this suicide classification system is in its ability to comprehensively identify suicidal events while limiting the over-identification of suicidal behavior.
Time Frame: Overall post Open-label Baseline treatment period (26 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Participants
  SI: Wish to be dead | 2
  SI: Non-specific active suicidal thoughts | 2
  SI: Any methods (not plan) without intent to act | 0
  SI: Some intent to act, without specific plan | 0
  SI: Specific plan and intent | 0
  SB: Preparatory acts or behavior | 0
  SB: Aborted attempt | 1
  SB: Interrupted attempt | 0
  SB: Actual attempt (non-fatal) | 0
  SB: Completed suicide | 0

4. Secondary Outcome: Time to Relapse During the 26-week Open-label Treatment Period for Subjects Who Demonstrated a Clinical Response to 4 Weeks of Treatment With SEP-363856
Description: Relapse is defined as the earliest occurrence of any of the following: - An increase in PANSS total score by ≥ 30% from the PANSS total score at clinical response and a CGI-S score ≥ 3; - Re-hospitalization for worsening of psychosis; - Emergence of suicidality, homicidality, and/or risk of harm to self or others.
Time Frame: From the time of clinical response to relapse or censor (one day after the last study drug dose)
Population: Relapse population, which includes subjects who received at least one dose of open-label treatment and demonstrated a clinical response to 4 weeks of treatment with SEP-363856. Clinical response is defined as meeting (1) a decrease in PANSS total score of ≥ 20% from double-blind Baseline, AND (2) a CGI-S score ≤ 4. For PBO-SEP subjects, clinical response was evaluated at Week 4 of study SEP361-201. For SEP-SEP subjects, clinical response was evaluated at Week 4 of study SEP361-202.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- PBO-SEP: Subjects who received Placebo in study SEP361-201 and SEP-363856 in study SEP361-202
- SEP-SEP: Subjects who received SEP-363856 in study SEP361-201 and SEP-363856 in study SEP361-202
Arm/Group | PBO-SEP | SEP-SEP
Number analyzed (Participants) | 59 | 51
Days | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events

5. Secondary Outcome: Rate of Relapse During the 26-week Open-label Treatment Period for Subjects Who Demonstrated a Clinical Response to 4 Weeks of Treatment With SEP-363856
Description: as for outcome 4
Time Frame: From the time of clinical response to relapse or censor (one day after the last study drug dose)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PBO-SEP | SEP-SEP
Number analyzed (Participants) | 59 | 51
Participants | 12 | 11

6. Secondary Outcome: Changes From Double-blind Baseline of Study SEP361-201 and Open-label Baseline of Study SEP361-202 in Positive and Negative Syndrome Scale (PANSS) Total Score and Subscale Scores (Positive, Negative, and General Psychopathology)
Description: PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210.
Time Frame: Double-blind Baseline (DB BLN), Open-label Baseline (OL BLN), Week 26 (Wk 26)
Population: Subjects with PANSS data missing at a particular time point did not contribute to the summary for that time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Units on a scale
  Total Score: DB BLN Observed | 101.5 (7.99)
  Total Score: OL BLN Observed | 83.1 (15.03)
  Total Score: Wk 26 Observed: number analyzed (Participants) | 104
  Total Score: Wk 26 Observed | 59.3 (12.45)
  Total Score: Chg from DB BLN at Wk 26: number analyzed (Participants) | 104
  Total Score: Chg from DB BLN at Wk 26 | -41.8 (13.98)
  Total Score: Chg from OL BLN at Wk 26: number analyzed (Participants) | 104
  Total Score: Chg from OL BLN at Wk 26 | -22.6 (15.48)
  Positive SS: DB BLN Observed | 25.7 (3.22)
  Positive SS: OL BLN Observed | 19.8 (4.96)
  Positive SS: Wk 26 Observed: number analyzed (Participants) | 104
  Positive SS: Wk 26 Observed | 12.2 (3.72)
  Positive SS: Chg from DB BLN at Wk 26: number analyzed (Participants) | 104
  Positive SS: Chg from DB BLN at Wk 26 | -13.5 (4.75)
  Positive SS: Chg from OL BLN at Wk 26: number analyzed (Participants) | 104
  Positive SS: Chg from OL BLN at Wk 26 | -7.3 (5.37)
  Negative SS: DB BLN Observed | 25.4 (4.03)
  Negative SS: OL BLN Observed | 22.3 (4.38)
  Negative SS: Wk 26 Observed: number analyzed (Participants) | 104
  Negative SS: Wk 26 Observed | 17.2 (4.10)
  Negative SS: Chg from DB BLN at Wk 26: number analyzed (Participants) | 104
  Negative SS: Chg from DB BLN at Wk 26 | -8.4 (4.48)
  Negative SS: Chg from OL BLN at Wk 26: number analyzed (Participants) | 104
  Negative SS: Chg from OL BLN at Wk 26 | -5.2 (4.20)
  Gen-Psychopathology SS: DB BLN Observed | 50.4 (5.01)
  Gen-Psychopathology SS: OL BLN Observed | 41.1 (7.93)
  Gen-Psychopathology SS: Wk 26 Observed: number analyzed (Participants) | 104
  Gen-Psychopathology SS: Wk 26 Observed | 30.0 (6.77)
  Gen-Psychopathology SS: Chg from DB BLN at Wk 26: number analyzed (Participants) | 104
  Gen-Psychopathology SS: Chg from DB BLN at Wk 26 | -19.9 (7.86)
  Gen-Psychopathology SS: Chg from OL BLN at Wk 26: number analyzed (Participants) | 104
  Gen-Psychopathology SS: Chg from OL BLN at Wk 26 | -10.2 (8.31)

7. Secondary Outcome: Change From Double-blind Baseline of Study SEP361-201 and Open-label Baseline of Study SEP361-202 in Clinical Global Impression - Severity (CGI-S) Score
Description: The CGI-S is a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.
Time Frame: Double-blind (DB) Baseline, Open-label (OL) Baseline, Week 26
Population: Subjects with CGI-S score data missing at a particular time point did not contribute to the summary for that time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Units on a scale
  CGI-S Score: DB Baseline Observed | 5.0 (0.42)
  CGI-S Score: OL Baseline Observed | 4.0 (0.84)
  CGI-S Score: Week 26 Observed: number analyzed (Participants) | 104
  CGI-S Score: Week 26 Observed | 3.0 (0.74)
  CGI-S Score: Change from DB Baseline at Week 26: number analyzed (Participants) | 104
  CGI-S Score: Change from DB Baseline at Week 26 | -2.0 (0.82)
  CGI-S Score: Change from OL Baseline at Week 26: number analyzed (Participants) | 104
  CGI-S Score: Change from OL Baseline at Week 26 | -1.0 (0.91)

8. Secondary Outcome: Change From Double-blind Baseline of Study SEP361-201 and Open-label Baseline of Study SEP361-202 in Brief Negative Symptom Scale (BNSS) Total Score
Description: The BNSS is a rating scale to measure the current level of severity of negative symptoms in schizophrenia and schizoaffective disorder. The measure is comprised of 13 individual items organized in 6 subscales. The 13 individual items provide a composite total score (ranging from 0 to 78). Each of the items are scored on a Likert-type 7-point scale from 0 - 6, where values of 0 indicates symptom is absent and a value of 6 means the symptom is a severe form.
Time Frame: Double-blind (DB) Baseline, Open-label (OL) Baseline, Week 26
Population: Subjects with BNSS total score data missing at a particular time point did not contribute to the summary for that time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Units on a scale
  Total Score: DB Baseline Observed: number analyzed (Participants) | 148
  Total Score: DB Baseline Observed | 38.4 (11.94)
  Total Score: OL Baseline Observed: number analyzed (Participants) | 150
  Total Score: OL Baseline Observed | 33.0 (11.41)
  Total Score: Week 26 Observed: number analyzed (Participants) | 104
  Total Score: Week 26 Observed | 22.5 (11.83)
  Total Score: Change from DB Baseline at Week 26: number analyzed (Participants) | 96
  Total Score: Change from DB Baseline at Week 26 | -16.8 (12.42)
  Total Score: Change from OL Baseline at Week 26: number analyzed (Participants) | 100
  Total Score: Change from OL Baseline at Week 26 | -11.3 (9.69)

9. Secondary Outcome: Change From Double-blind Baseline of Study SEP361-201 and Open-label Baseline of Study SEP361-202 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts. Each item is scored in a range of 0 to 6 points, with higher scores indicating increased depressive symptoms.
  Total score will be equal to the sum of the 10 items (range between 0 and 60).
Time Frame: Double-blind (DB) Baseline, Open-label (OL) Baseline, Week 26
Population: Subjects with MADRS total score data missing at a particular time point did not contribute to the summary for that time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SEP-363856
Number analyzed (Participants) | 156
Units on a scale
  Total Score: DB Baseline Observed | 12.6 (7.25)
  Total Score: OL Baseline Observed | 9.2 (6.33)
  Total Score: Week 26 Observed: number analyzed (Participants) | 104
  Total Score: Week 26 Observed | 4.4 (4.72)
  Total Score: Change from DB Baseline at Week 26: number analyzed (Participants) | 104
  Total Score: Change from DB Baseline at Week 26 | -8.1 (6.44)
  Total Score: Change from OL Baseline at Week 26: number analyzed (Participants) | 104
  Total Score: Change from OL Baseline at Week 26 | -4.5 (5.28)

10. Secondary Outcome: Proportion of Subjects Who Achieved a Response, Defined as a 20% or Greater Improvement in Positive and Negative Syndrome Scale (PANSS) Total Score From Double-blind Baseline of Study SEP361-201
Description: as for outcome 6
Time Frame: Week 26
Population: Subjects who received at least one dose of open-label treatment and had PANSS total score data available at Double-blind Baseline and Week 26 are included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PBO-SEP | SEP-SEP
Number analyzed (Participants) | 53 | 51
Participants | 52 | 49

ADVERSE EVENTS:
Time Frame: From first dose of study drug to last study visit (27 weeks)
Arm/Group | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 15/156
Other Adverse Events (participants affected / at risk) | 39/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-363856 (N=156)
Acute psychosis (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 11 (11)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-363856 (N=156)
Headache (Nervous system disorders) | 18 (36)
Anxiety (Psychiatric disorders) | 8 (36)
Insomnia (Psychiatric disorders) | 13 (24)
Schizophrenia (Psychiatric disorders) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT02970929/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02970929/SAP_001.pdf